CLINICAL TRIAL: NCT07395232
Title: A Phase 3, Multicenter, Randomized, Double-Masked, Vehicle-Controlled Study to Demonstrate Efficacy and Safety of DFL24498 Eye Drop Solution in Adult Participants With Atopic Keratoconjunctivitis (AKC)
Brief Title: An Efficacy and Safety Study of DFL24498 in the Treatment of AKC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICY-AKC-301; 2025-522291-83-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-22; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Atopic Keratoconjunctivitis
Keywords: chronic, recurrent ocular surface inflammation,; Atopic Keratoconjunctivitis; DFL24498; Ophthalmic solution; Vehicle controlled; Eye drop solution; Corneal involvement
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — dexamethasone 21-phosphate; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DFL24498 (Experimental): Participants will be administered with DFL24498 eye drops in both eyes.
  Interventions: Drug: DFL24498; Drug: dexamethasone sodium phosphate (DSP) ophthalmic solution
- Vehicle (Placebo Comparator): Participants will be administered with vehicle eye drops in both eyes.
  Interventions: Drug: Vehicle; Drug: dexamethasone sodium phosphate (DSP) ophthalmic solution

INTERVENTIONS:
Drug: DFL24498 — DFL24498 will be instilled in each eye for 12 Weeks.
  Arms: DFL24498
Drug: Vehicle — Vehicle eye drops without active drug will be instilled in each eye for 12 Weeks.
  Arms: Vehicle
Drug: dexamethasone sodium phosphate (DSP) ophthalmic solution — Rescue medication may be administered as required at the Investigator discretion.

SUMMARY:
This is a phase 3, multicenter, randomized, double-masked, parallel-group, vehicle-controlled study to evaluate the safety and efficacy of DFL24498 compared with vehicle ophthalmic solution, in participants with AKC. Approximately 138 participants who meet all eligibility criteria will be enrolled in the study.

DETAILED DESCRIPTION:
The study will consist of 3 periods:

1. Screening period (from Day -7 ± 1 to Day 1),
2. Treatment Period (from randomization through Week12) and
3. Follow-up period (Weeks 13 to 16).

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Men or women aged ≥ 18 and ≤ 65 years of age.
2. Diagnosis of AKC in both eyes, including the presence or medical history of the following:

   1. other atopic condition (ie,. atopic dermatitis, periocular eczema, asthma, allergic rhinitis), AND
   2. chronic allergic blepharoconjunctivitis and/or keratoconjunctivitis.
3. Ocular itching of at least 50 as assessed by VAS scale.
4. Corneal fluorescein staining assessed by modified Oxford scale of at least grade 1 AND a bulbar conjunctival hyperemia assessed by VBR 10 scale of at least 40 (range 0 to 100) in the same eye.
5. A composite symptoms score (CSyS) ≥ 5 (sum of the severity scores graded 0 to 3 for each of the following: itching, tearing, ocular discomfort, photophobia, and mucous discharge score) (CSyS range of 0 to 15).
6. If a woman of childbearing potential (WOCBP), must have a negative pregnancy test at both screening and baseline visit, and use an acceptable contraception method.

Exclusion Criteria:

Participants will be excluded if any of the following criteria apply:

1. Inability to speak and understand the local language sufficiently to understand the nature of the study, to provide written informed consent, and to allow the completion of all study assessments.
2. Evidence of an active ocular infection in either eye.
3. Intraocular inflammation defined as anterior chamber flare > 0 by Standardization of Uveitis Nomenclature (SUN) grading, in either eye.
4. Known or suspected ocular malignancy (ocular surface, intraocular, ocular adnexa).
5. Presence of cancer or any other systemic or unstable disease that may affect the ability to participate in the clinical study in the opinion of the investigator including basal cell carcinoma.
6. Participants that are anatomically monocular.
7. Systemic disease not stabilized within 1 month before the screening visit (eg, diabetes with glycemia out of range, thyroid malfunction) or judged by the investigator to be incompatible with the study (eg, current systemic infections) or with a condition incompatible with the frequent assessment required by the study.

Note: Additional protocol defined Inclusion/Exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline at week 6 in ocular itching score assessed by visual analog scale (VAS). | Baseline and at Week 6
  The ocular itching VAS ranges from 0 to 100 mm (0 mm = no ocular itching at all, 100 mm = intolerable itching). Participants will be asked to subjectively rate the current severity of ocular itching at each time point.

SECONDARY OUTCOMES:
Change from baseline at week 6 in corneal epithelial fluorescein staining, scored by modified Oxford scale, in the study eye. | Baseline and at Week 6
  Fluorescein will be applied to the inferior fornix of the palpebral conjunctiva of each eye. To avoid the phenomenon of quenching, staining will be assessed within 1 to 4 minutes from fluorescein instillation. Examination will be performed at the slit-lamp using blue (cobalt) light. Corneal fluorescein staining will be graded according to the modified Oxford scale (7-point scale: 0, 0.5. 1, 2, 3, 4, 5).
Change from baseline at week 6 in bulbar conjunctival hyperemia assessed by Validated Bulbar Redness (VBR) 10 scale (0 to 100), in the study eye. | Baseline and at Week 6
  Bulbar conjunctival redness will be assessed at the slit-lamp examination using white light prior to vital dye instillation and graded according to the VBR 10 scale.
Change from baseline over time in ocular itching score assessed by VAS. | Baseline and at Week 4, Week 6, Week 8, Week 12, and Week 16
  The ocular itching VAS ranges from 0 to 100 mm (0 mm = no ocular itching at all, 100 mm = intolerable itching). Participants will be asked to subjectively rate the current severity of ocular itching at each time point.
Change from baseline over time in ocular symptoms of itching, tearing, discomfort, mucous discharge, and photophobia on a 4-point scale (0 to 3). | Baseline and at Week 4, Week 6, Week 8, Week 12, and Week 16
  Ocular symptoms are assessed using a 4-point severity scale ranging from 0 (none) to 3 (severe). Five ocular symptoms, itching, tearing, ocular discomfort (including burning, stinging, and foreign body sensation), mucous discharge, and photophobia are evaluated in the study eye. A composite symptom score is described in calculated at screening and Baseline by summing the individual symptom scores, resulting in a total score range of 0 to 15, with higher scores indicating greater symptom severity.
Change from baseline over time in corneal fluorescein staining (modified Oxford scale) in the study eye. | Baseline and at Week 4, Week 6, Week 8, Week 12, and Week 16
  Corneal fluorescein staining modified Oxford scale (0-5) as per corneal dot count in each eye.
Change from baseline over time in bulbar conjunctival hyperemia assessed by VBR 10 scale (0 to 100) in the study eye. | Baseline and at Week 4, Week 6, Week 8, Week 12, and Week 16
  Bulbar conjunctival hyperemia assessed by Validated Bulbar Redness (VBR) 10 scale (0 to 100).
Change from baseline over time in signs of tarsal papillary reaction, corneal neovascularization, cicatrizing conjunctivitis and blepharitis on a 4-point scale (0 to 3) in the study eye. | Baseline and at Week 4, Week 6, Week 8, Week 12, and Week 16
  Change in signs on a 4-point scale (0 to 3) in the study eye.
Change from baseline at week 6 and 12 in the QoL scores assessed by the Standardized Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ-S) | Baseline and at Week 6 and Week 12.
  Standardized Rhinoconjunctivitis QoL Questionnaire (RQLQ[S]) is a validated questionnaire that assesses QoL specifically in patients with rhinoconjunctivitis. There are 28 questions, which are categorized under 7 domains (activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional). Each question is scored on a 7-point scale from no impairment (score 0) to severe impairment (score 6).
Patient Global Impression of Change (PGIC) at week 6 and week 12. | At week 6 and week 12.
  PGIC is a short questionnaire used to assess how a participant perceives changes in their condition following treatment, on a scale ranging from 1 to 7.
Number of Participants receiving rescue medication over time after week 6 | Week 6 to Week 12
  Participants who received rescued medication over time after week 6 (visit 4).
Number of participants with treatment-emergent adverse events and serious adverse events (SAEs) | Up to Week 16
  Any adverse events occurring or worsening after the first administration of investigational product is classified as "treatment-emergent" adverse events and does not necessarily have a causal relationship with the intervention. A SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product, and is medically important.
Change from baseline over time in best corrected distance visual acuity (BCDVA) in each eye. | Baseline and at Week 4, Week 6, Week 8, Week 12, and Week 16
  Best corrected visual acuity (BCDVA) is determined by careful refraction according to the standard protocol for refraction. BCDVA is measured by Early Treatment of Diabetic Retinopathy Study chart.
Change from baseline at week 12 in corneal endothelial cell density in each eye (only at selected sites that have the required equipment). | Baseline and at week 12
  Corneal central region endothelial cell density will be determined for each eye using specular microscopy and expressed as the number of cells/mm2 using the Cell Density readout provided by the software.
Change from baseline at week 12 in dilated fundus exam in each eye (proportion of participants with vitritis, retinal or vitreal hemorrhages, increase in cup-to-disc ratio, retinal or posterior vitreal detachment, retinal tears, or maculopathy). | Baseline and at week 12
  After specular microscopy, mydriatic drops will be instilled in both eyes and once adequate dilation is achieved, a fundal exam shall be performed to examine the vitreous, retina, and optic nerve.
Change from baseline over time in intraocular pressure in each eye. | Baseline and at Week 6 and Week 12
  IOP will be assessed by applanation tonometry for each eye and will be measured in mmHg.
Number of participants discontinued due to tolerability during the treatment period | Baseline to week 12
  Treatment discontinuation rate due to tolerability.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (8):
  - Bowden Eye Associates - Southside Location, Jacksonville, Florida
  - University of Miami, Miller School of Medicine, Bascom Palmer Eye Institute, Miami, Florida
  - Clayton Eye Clinical Research, Morrow, Georgia
  - Ophthalmology Associates, St Louis, Missouri
  - NYU Langone Health - Eye Center, New York, New York
  - Duke Eye Center - Ophthalmology, Durham, North Carolina
  - Total Eye Care, PA, Memphis, Tennessee
  - Baylor University Jamail Specialty Care Center- Alkek Eye Center- Ophthalmology, Houston, Texas
- Italy (6):
  - IRCCS AOU di Bologna - Policlinico Sant'Orsola UO Oftalmologia, Bologna
  - Ospedale SS Annunziata, ASL 2 Lanciano Vasto Chieti, Chieti
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma
  - AOU Policlinico Umberto I, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Spain (5):
  - METAVISION ARRUZAFA S.L. (Hospital Arruzafa), Córdoba
  - Miranza Galicia, Santiago de Compostela
  - Fundación de Oftalmología Médica de la Comunitat Valenciana (FOM), Valencia
  - OBA - Universidad de Valladolid, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No